CLINICAL TRIAL: NCT06561594
Title: A Multicenter, Randomized, Double-blind, Phase III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Human Follicle-stimulating Hormone-CTP Fusion Protein Injection or Placebo Combined With Chorionic Gonadotropin for Injection in Idiopathic Hypogonadotropin Hypogonadism
Brief Title: To Evaluate Recombinant Human Follicle Stimulating Hormone-CTP Fusion Protein Injection or Placebo Combined With Chorionic Gonadotropin for Injection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci094-303
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism

STUDY DESIGN:
Intervention Model Description: recombinant human follicle-stimulating hormone-CTP Fusion protein injection or placebo combined with chorionic gonadotropin for injection
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 30subjects：GenSci094 was administered for 12 weeks，150ug/0.5ml（weight>60kg）or 100ug/0.5ml（weight≤60kg）；GenSci094 with chorionic gonadotropin for injection was administered for 52 weeks，150ug/0.5ml（weight>60kg）or 100ug/0.5ml（weight≤60kg）with chorionic gonadotropin for injection.
  Interventions: Drug: recombinant human follicle-stimulating hormone-CTP Fusion protein injection
- Placebo group (Placebo Comparator): 30subjects：GenSci094 Placebo was administered for 12 weeks，150ug/0.5ml（weight≥60kg）or 100ug/0.5ml（weight<60kg）；GenSci094 Placebo with chorionic gonadotropin for injection was administered for 52 weeks，150ug/0.5ml（weight≥60kg）or 100ug/0.5ml（weight<60kg）with chorionic gonadotropin for injection.
  Interventions: Drug: recombinant human follicle-stimulating hormone-CTP Fusion protein injection Placebo

INTERVENTIONS:
Drug: recombinant human follicle-stimulating hormone-CTP Fusion protein injection — IF Weight > 60kg，150ug, H. Administer the drug once every 14 days for 64 weeks；IF Weight >≤60kg，100ug, H. Administer the drug once every 14 days for 64 weeks
  Arms: Experimental group
Drug: recombinant human follicle-stimulating hormone-CTP Fusion protein injection Placebo — 0.5ml, H. Administer the drug once every 14 days for 64 weeks
  Arms: Placebo group

SUMMARY:
This study was conducted to evaluate recombinant human follicle stimulating hormone-CTP fusion protein injection or placebo combined with chorionic gonadotropin for injection

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, Phase III clinical study to evaluate the efficacy and safety of recombinant human follicle-stimulating hormone-CTP Fusion protein injection or placebo combined with chorionic gonadotropin for injection to initiate or restore puberty in idiopathic hypogonadotropin hypogonadism in adolescent males aged 14 to 18 years.

ELIGIBILITY:
Inclusion Criteria:

* The guardian and subject are aware of the study procedures, available alternative treatments, and the risks of participating in the study, and voluntarily sign a written ICF to voluntarily participate in the study.
* Age 14-18 years old (excluding 18 years old) at the time of signing the ICF, with bone age greater than 12 years old.
* Height ≥145cm and body mass index (BMI) < 30kg/m2 when signing ICF.
* Diagnosis of idiopathic or congenital hypogonadotropic hypogonadism.
* The presence of bilateral pre-gonadal onset testis during the screening period: testicular volume <4 mL on each side (determined by ultrasound and evaluated by 2 qualified ultrasound specialists authorized by the researchers of the research center).
* The circulating gonadotropin (Gn) level was low (FSH≤1 IU/L and LH≤1 IU/L) during the screening period, and the peak LH value of GnRH excitation test was ≤4 IU/L.
* Serum testosterone T ≤ 1 ng/mL during the screening period.
* The normal range of other pituitary hormones during the screening period (judged by the researcher).
* Lesions detected by MRI on the head within 3 months before or during screening were normal or determined by the investigator to have no impact on the study.
* Consent to the use of reliable contraception (e.g. abstinence, condoms, etc.) by yourself and your sexual partner during the study period and for 3 months after the study drug treatment.

Exclusion Criteria:

There is primary hypogonadism (e.g., Klinefelter syndrome).

* Hypogonadotropic hypogonadism caused by tumor, surgery, trauma, infection, or immune factors in the hypothalamic sella or pituitary gland.
* History of unilateral or bilateral cryptorchidism and the presence of clinically significant testicular lesions (orchitis, testicular tumor, testicular torsion, severe varicocele (grade III), testicular atrophy, obstructive azoospermia, etc.).
* Researchers identified uncontrolled endocrine diseases, including thyroid, adrenal diseases, diabetes, etc.
* History of malignant tumors within 5 years prior to the screening period.
* Patients who have received GnRH, gonadotropin or oral androgen (testosterone, etc.) therapy within 1 month before signing ICF, or who have received testosterone undecanoate intramuscular injection therapy within 1 year before signing ICF.
* History of drug or substance abuse within 1 year prior to signing the ICF, drugs known to impair testicular function or affect the production of sex hormones, or alcohol abuse.
* Abnormal liver and kidney function during screening, i.e. liver function: alanine aminotransferase and/or aspartate aminotransferase higher than 2 times the upper limit of normal (>2×Upper limit of normal); Renal function: Creatinine and/or urea/urea nitrogen are 2 times higher than the upper limit of normal (>2×Upper limit of normal).
* During the screening period, patients with systemic diseases (such as metabolic abnormalities, circulatory, digestive, nervous system, etc.) judged by the researchers are not suitable for participation in this study.
* Current thromboembolic disease or known prior history.
* Hepatitis B surface antigen, hepatitis C antibody, HIV antibody and treponema pallidum antibody positive.●
* People who are allergic to the active ingredients or excipients of FSH and hCG drugs or have a history of related allergies, or have a clear contraindication of drug use.
* Participants who participated in other interventional clinical trials and used experimental drugs within 3 months prior to screening.
* Patients with a history of depression or mental disorders.
* Due to risk considerations, the researchers did not consider it appropriate to participate in other situations in this study.

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2024-11-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in testicular volume (the sum of the volumes of the left and right testes measured on ultrasonography) after 64 weeks | 64 weeks after administration

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Anhui Children's Hospital, Hefei, Anhui
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Women and Children's Medical Center Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Jiangxi Children's Hospital, Nanchang, Jiangxi
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Jining Medical College, Jining, Shangdong
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Pediatric Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women and Children's Central Hospital, Chengdu, Sichuan